CLINICAL TRIAL: NCT04902651
Title: A PROSPECTIVE, CONTROLLED, RANDOMIZED, OPEN-LABEL PREMARKET MULTICENTER STUDY OF THE PERFORMANCE OF THE HM242-GEL VS COMPARATOR IN PATIENTS UNDER THE CONDITION OF VENOUS LEG ULCER
Brief Title: HM242-Gel vs Comparator
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: stopped for futility
Sponsor: B. Braun Ltd. Centre of Excellence Infection Control (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPM-G-H-2004
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2021-05

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HM242-Gel (Experimental)
  Interventions: Device: HM242-Gel
- Intrasite Gel (Active Comparator)
  Interventions: Device: Intrasite Gel

INTERVENTIONS:
Device: HM242-Gel — HM242-Gel compared to Intrasite Gel in patients with a venous leg ulcer
  Arms: HM242-Gel
Device: Intrasite Gel — HM242-Gel compared to Intrasite Gel in patients with a venous leg ulcer
  Arms: Intrasite Gel

SUMMARY:
The primary objective of the study is to demonstrate that the HM242-Gel performs at least comparably to INTRASITE Gel with regard to wound healing.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of at least 18 years at the time of enrolment
2. The legal capacity and ability to understand the nature, risks, significance and scope of the clinical trial and to determine his or her will accordingly
3. Signed form of consent, including the understanding of and willingness by the patient to participate in the clinical study and ability to comply with study procedures and study visit schedule
4. Patients must be willing to have all dressing changes performed by the wound specialist, with no treatments at home
5. Presence of at least one venous ulcer of the lower leg extending through the full thickness of the skin but not down to muscle, tendon or bone
6. Size of study ulcer ≥ 2cm² and ≤ 100cm² measured using the tracing method.
7. Presence of venous leg ulcer for at least 6 weeks, but not longer than 12 months
8. Ankle Brachial Pressure Index (ABI) > 0.75
9. In the case of a female patient of childbearing potential, willingness to use highly effective methods of contraception (failure rate of < 1% when used consistently and correctly);acceptable contraceptive measures in this trial are: combined pill and progestin-only pill, contraceptive patch, ring or injection, Etonogestrel implant, intrauterine device (IUD) (copper and Levonogestrel), male sterilization (vasectomy), female sterilization (abdominal, laparoscopic, hysteroscopic), or sexual abstinence.

Exclusion Criteria:

1. Patients kept in an institution due to an official or court order
2. Patients dependent on the Sponsor, Investigator or Site
3. Patients suspected of having SARS-CoV-2 infection or COVID-19 disease
4. Study ulcer judged by the Investigator to be caused by a medical condition other than venous insufficiency
5. Study ulcer with signs and symptoms of infection, or under suspicion of cancer
6. Study ulcer under treatment with topical antimicrobials within past two weeks or systemic antimicrobial treatment within past two weeks
7. In the case of heavily exuding ulcers, if in the opinion of Investigator the patient is not suitable for treatment with gel
8. More than two venous leg ulcers or more than two chronic wounds
9. Dementia stage greater than 3 according to Reisberg
10. Known allergies against wound dressings used in the study
11. Known chronical skin diseases, dermatoses, or known allergies or other conditions which might trigger dermatitis
12. Acute cases of substance use disorders (ICD-10 F1x.1 or F1x.2)
13. Buerger's disease
14. Participation in Medical Device trials less than 4 weeks ago or participation in Drug trials less than six months ago
15. Terminally ill patients
16. Patients with poorly managed diabetes mellitus: absence of a glycated hemoglobin test within the last 3 months or a result of HbA1c ≥ 8% not older than 3 months, or a major diabetes-related incident within the past 4 weeks
17. Ulcers of diabetic origin
18. Patients under treatment with systemic corticosteroids, immunosuppressant, cytotoxic chemotherapy, or radiotherapy
19. Presence of one or more medical conditions (other than venous insufficiency and diabetes) as determined by medical history, which:

    * Is known to interfere with the wound healing process (e.g. arteriopathy, vasculitis, rheumatoid arthritis, systemic lupus erythematosus, other auto-immune diseases, cancer, immunodeficiency, severe lymphedema of the leg, thrombophilia)
    * In the opinion of the Investigator, would make the patient an inappropriate candidate for this venous ulcer healing study (e.g. malnutrition, hygiene, obesity)
20. Pregnant or lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to demonstrate that the HM242-Gel performs at least comparably to INTRASITE Gel with regard to wound healing. | 28 days
  The primary variable is defined as the relative reduction of the wound area of a patient in percentage 28 days (4 weeks) after baseline. The wound size area is measured on site by the tracing method.

CONTACTS AND LOCATIONS:
Locations (3):
- Kožní ambulance Fialová, s.r.o., Prague, Praha 6, Czechia
- Slovakia (2):
  - Viliam Cibik, Pruské
  - Rudolf Suchy, Trenčín

IPD SHARING:
Plan to Share IPD: No